CLINICAL TRIAL: NCT05392608
Title: SEQUence of Endocrine Therapy in Advanced Luminal Breast Cancer (SEQUEL-Breast): A Phase 2 Study on Fulvestrant Beyond Progression in Combination With Alpelisib for PIK3CA-mutated, Hormone-receptor Positive HER2 Negative Advanced Breast Cancer
Brief Title: SEQUence of Endocrine Therapy in Advanced Luminal Breast Cancer (SEQUEL-Breast)
Acronym: SEQUEL-Breast
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Borstkanker Onderzoek Groep (Network)
Collaborators: Novartis Pharma B.V. (Unknown); BOOG Study Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BOOG 2021-01 SEQUEL-Breast
Record Dates: First submitted 2022-05-16; First posted 2022-05-26 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Neoplasm, Breast; Congenital, Familial and Genetic Disorders
Keywords: Hormone receptor positive HER2 negative breast cancer; PIK3CA-activated mutation
MeSH Terms: conditions — Breast Neoplasms; Genetic Diseases, Inborn | interventions — Alpelisib; Tablets; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm A (one-arm study) (Experimental): Alpelisib plus fulvestrant beyond progression
  Interventions: Drug: Alpelisib 150 MG Oral Tablet [Piqray]; Drug: Fulvestrant

INTERVENTIONS:
Drug: Alpelisib 150 MG Oral Tablet [Piqray] — Alpelisib 300mg once daily (may be reduced to 1dd250 or 1dd200mg in case of toxicity)
  Other Names: Piqray
Drug: Fulvestrant — Fulvestrant 300mg 1x/four weeks
  Other Names: Faslodex

SUMMARY:
The study is a nationwide, multicenter single-arm phase 2 study. The current phase 2 study investigates the efficacy of the combination of fulvestrant and alpelisib directly after progression on fulvestrant (either in first or second line, with or without previous use of CDK4/6-inhibitor) in patients with HR+ HER2- advanced breast cancer with PIK3CA mutated tumors.

All eligible patients must have progressive disease on fulvestrant as latest treatment line.

Previous treatment with a CDK4/6 inhibitor in first or second line is obligatory. After progressive disease is confirmed, it is important to continue fulvestrant (without CDK4/6 inhibition) during the screening period awaiting study enrollment.

After study enrollment all participants will be treated with alpelisib and fulvestrant beyond progression. Follow-up time will be until progression or death or until a different oncolytic treatment has started (in case no progressive disease during previous fulvestrant and alpelisib treatment has been documented).

Should participants discontinue due to reasons other than progression or death (e.g. toxicity), then they should still be evaluated for disease progression every 8 weeks as per protocol until progression, unless they do not wish to proceed with these screenings, or receive a different oncolytic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult women and men (≥ 18 years of age) with proven diagnosis of adenocarcino-ma of the breast withlocoregional recurrent or metastatic disease not amenable to resection or radiation therapy with curative intent andfor whom chemotherapy is not clinically indicated
* Estrogen receptor (ER) expression >10% and/or progesterone receptor (PR) expression >10% breast cancerbased on local la-boratory results. Tumor must be HER2- as defined by ASCO-CAP guidelines
* Patients must have progressed on fulvestrant as a preceding treatment line (as first or second line therapy)
* Previous treatment with a CDK4/6 inhibitor in the advanced setting
* The presence of an activating PIK3CA mutation
* Evaluable disease* as defined per RECIST v.1.1
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2

Exclusion Criteria:

* Patients with advanced, symptomatic, visceral spread, who are at risk of life-threatening complications in theshort term
* Known active uncontrolled or symptomatic CNS metastases, carcinomatous meningitis, or leptomeningealdisease as indicated by clinical symptoms, cerebral edema, and/or progressive growth
* Prior treatment with a PI3K /AKT/mTOR inhibitor
* Type 1 diabetes or uncontrolled type 2 diabetes (Hba1C > 68 mmol/mol)
* Clinically significant, uncontrolled heart disease and/or recent cardiac events

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-06-02 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From registration to progression, assessed up to 36 months
  Defined as time from study enrollment to disease progression or death from any cause, with censoring when fulvestrant and alpelisib are stopped and another treatment is initiated without confirmed disease progression.

SECONDARY OUTCOMES:
'On treatment' Progression-free survival (PFS) | From registration to progression, assessed up to 36 months
  Defined as time from study enrollment to disease progression or death from any cause, with censoring when fulvestrant and alpelisib are stopped earlier than disease progression
Objective Response Rate | From registration to progression, assessed up to 36 months
  Described as complete response (CR) or partial response (PR)
Clinical Benefit Rate | From registration to progression, assessed up to 36 months
  Described as stable disease (SD), PR, or CR
Duration of Response (DoR) | From registration to progression, assessed up to 36 months
  Duration of Response

OTHER OUTCOMES:
Determine circulating tumor DNA (ctDNA) in plasma before and during treatment | At baseline, 2 weeks of treatment, 8 weeks of treatment and every 8 weeks until disease progression. Assessed up to 36 months
  Exploratory endpoint; determine circulating tumor DNA (ctDNA) in plasma before and during treatment, to investigate the prognostic and possibly predictive values of these measures

CONTACTS AND LOCATIONS:
Overall Officials: Vincent V.O. Dezentjé, MD PhD, Principal Investigator — NKI-AvL; Inge I.R. Konings, MD PhD, Principal Investigator — Amsterdam UMC; Monique M.E.M.M. Bos, MD PhD, Principal Investigator — Erasmuc MC
Locations (25):
- Netherlands (25):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Ziekenhuisgroep Twente, Almelo
  - Meander Medisch Centrum, Amersfoort
  - Ziekenhuis Amstelland, Amstelveen
  - Amsterdam UMC, Amsterdam
  - Antoni van Leeuwenhoek, Amsterdam
  - Gelre Ziekenhuizen, Apeldoorn
  - Rijnstate, Arnhem
  - Amphia, Breda
  - Reinier de Graaf Gasthuis, Delft
  - Deventer ziekenhuis, Deventer
  - Máxima Medisch Centrum, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - Admiraal de Ruyter Ziekenhuis, Goes
  - Martini Ziekenhuis, Groningen
  - Spaarne Gasthuis, Hoofddorp
  - Medisch Centrum Leeuwarden, Leeuwarden
  - St. Antonius Ziekenhuis, Nieuwegein
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Maasstad Ziekenhuis, Rotterdam
  - Franciscus Gasthuis & Vlietland, Schiedam
  - HagaZiekenhuis, The Hague
  - Elisabeth-TweeSteden Ziekenhuis, Tilburg
  - VieCuri Medisch Centrum, Venlo

IPD SHARING:
Plan to Share IPD: No